CLINICAL TRIAL: NCT04768998
Title: Intersectoral Platform (SÜP) of the National Pandemic Cohort Network (NAPKON)
Acronym: SUEP-NAPKON
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Goethe University (Other)
Collaborators: Nationwide Network of University Medicine (NUM) on Covid-19 (Unknown)
Responsible Party: Principal Investigator, Janne Vehreschild, Prof. Dr. med, Goethe University
Other Study IDs: 01KX2021
Record Dates: First submitted 2021-01-15; First posted 2021-02-24 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2)
Keywords: SARS-CoV-2; COVID-19; Coronavirus; Cohort; NAPKON; NAPKON-SÜP; Quality of life; longterm morbidity
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, respiratory samples (nose and throat swab, endotracheal aspirate, nasopharyngeal aspirate), urine
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Intersectoral Platform (SÜP) of the National Pandemic Cohort Network (NAPKON): Streamlined sampling of biomaterials and core data elements (GErman Corona COnsensus data set GECOO), with other NAPKON study platforms (HAP, POP).
  Interventions: Other: Observational of different courses of SARS-CoV-2 infection in different phases (acute vs. post-acute) and settings
- Populationbased Platform (POP) of the National Pandemic Cohort Network (NAPKON): Streamlined sampling of biomaterials and core data elements (GErman Corona COnsensus data set GECOO), with other NAPKON study platforms (HAP, SUEP).
  Interventions: Other: Observational of different courses of SARS-CoV-2 infection in different phases (acute vs. post-acute) and settings
- High-Resolution Platform (HAP) of the National Pandemic Cohort Network (NAPKON): Streamlined sampling of biomaterials and core data elements (GErman Corona COnsensus data set GECOO), with other NAPKON study platforms (POP, SUEP).
  Interventions: Other: Observational of different courses of SARS-CoV-2 infection in different phases (acute vs. post-acute) and settings

INTERVENTIONS:
Other: Observational of different courses of SARS-CoV-2 infection in different phases (acute vs. post-acute) and settings — Observatory Cohorts focusing (I) on subjects after SARS-CoV-2 infection that are recruited from the general population (POP), and on subjects with acute SARS-CoV-2 infections recruited (II) in university hospital high-care settings or (III) general health care.

SUMMARY:
The intersectoral platform is part of the National Pandemic Cohort Network (NAPKON) and will be used to provide a comprehensive and harmonized collection of data and biomaterial for researchers from national consortia, pharmaceutical companies and for participation in international research collaborations for the purpose of studying COVID-19 disease and future pandemics.

DETAILED DESCRIPTION:
The intersectoral platform is part of the National Pandemic Cohort Network (NAPKON), which, together and in interaction with other components of the National Research Network of University Medicine on COVID-19 (NUM), provides the essential basis for the successful understanding and thus combating pandemics using the example of coronavirus disease 2019 (COVID-19). NAPKON represents a sustainable, integrative and comprehensive concept that provides benefits for society as a whole in defending against and coping with pandemics, especially at the level of public health care, in hospital and patient management and from the individual patient's perspective.

The intersectoral platform records data and biomaterial of severe acute respiratory syndrome coronavirus type 2 (SARS-CoV-2)-infected patients through a network of university clinics, hospitals at all levels of care, general practitioners and specialist practices with appropriate study experience and infrastructure. The longitudinal phenotyping programme tracks patients for up to one year and collects detailed and harmonized clinical data as well as biomaterial. Follow-up data is enriched by patient-reported outcomes (PROM) and recruitment is intensified by focusing on hot-spot regions. Mobile study teams are used to reach, among others, long-term care and rehabilitation facilities, thus mapping all structural elements of the German care network.

The primary aim of the intersectoral platform is to provide a comprehensive and harmonized collection of data and biomaterial for researchers from national consortia, pharmaceutical companies and for participation in international research collaborations for the purpose of studying COVID-19 disease and future pandemics.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Compliance with the case definition (a-c):

   1. Polymerase chain reaction (PCR) or rapid test diagnosis from nasopharynx, bronchoalveolar lavage, oropharynx, stool and/or blood
   2. or a combination of:

      * negative molecular detection of SARS-CoV-2 AND
      * characteristic radiological findings AND
      * respiratory tract infection AND
      * absence of a more likely cause of disease, in particular other chronic lung diseases AND
      * Negative test for influenza
   3. or (control group) a combination of:

      * negative molecular detection of SARS-CoV-2 AND
      * respiratory tract infection AND
      * absence of a more likely cause of disease, in particular other chronic lung diseases AND
      * attempt of pathogen identification from respiratory material with at least culture and influenza test
3. The baseline visit needs to be performed a maximum of 7 days (168h) after sampling and 4 days (96h) after the case definition is available.
4. Signed informed consent

Exclusion Criteria:

1. Age <18 years
2. Paediatric patients will not be included at the beginning of the study (amendment in preparation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enrol eligible patients (in- and outpatients) with confirmed SARS-CoV-2 infection.
  Data and biospecimens will be collected during predefined study visits and patients are monitored up to 12 months after diagnosis.
Sampling Method: Probability Sample
Enrollment: 6550 (Estimated)
Dates: Start 2020-11-04 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Longitudinal collection of data and biomaterial | day 1 of enrollment in the study, immediately before discharge, 3 and 12 months after diagnosis
  To provide a comprehensive and harmonised collection of data and biomaterial for researchers from national consortia, pharmaceutical companies and for participation in international research collaborations for the purpose of studying COVID-19 and future pandemics.

SECONDARY OUTCOMES:
Number of cases of SARS-CoV-2 infection | 12 months
  Determine the number of cases of SARS-CoV-2 according to:
  * Severity of the disease
  * Deaths
  * Treatment status
  * Lengths of hospitalization
  * Duration of oxygen therapy
  * Underlying disease
Changes in concentration of inflammatory parameters. | Assessement at each study visit until discharge or death, assessed up to 12 months
  The changes of inflammatory parameters such as C-reactive protein (CRP) [mg/l], will be recorded and evaluated at all visits during the acute phase, if provided.
Changes in concentration of cardiac parameters. | Assessement at each study visit until discharge or death, assessed up to 12 months
  The changes of Fibrinogen [µmol/l] will be recorded and evaluated at all visits during the acute phase, if provided.
Changes in concentration of urine parameters. | Assessment of the urine parameters will be performed at all visits during the acute phase until discharge or death, assessed up to 12 months
  The changes in concentration of urine parameters such as Albumine ([mg/g Creatinin], will be recorded and evaluated, if provided.
Changes in Patient-reported Quality of life recorded with the help of the European Quality of Life 5 Dimensions 5 Level Version (Eq5d5l) questionnaire. | Date of admission, immediately before discharge, 3, 6, 12 months after first diagnosis
  Health related quality of life after hospital discharge will be assessed with the questionnaire European Quality of Life 5 Dimensions 5 Level Version (Eq5d5l)
Changes in body temperature. | Assessement at each study visit until discharge or death, assessed up to 12 months
  Assessment of the patient´s body temperature will be performed at all visits during the acute phase.
Changes in blood pressure. | Assessement at each study visit until discharge or death, assessed up to 12 months
  Assessment of the patient´s blood pressure will be performed at all visits during the acute phase.
Changes in heart rate. | Assessement at each study visit until discharge or death, assessed up to 12 months
  Assessment of the patient´s heart rate will be performed at all visits during the acute phase.
Changes in breath frequency. | Assessement at each study visit until discharge or death, assessed up to 12 months
  Assessment of the patient´s breath frequency will be performed at all visits during the acute phase.
Changes in peripheral oxygen saturation. | Assessement at each study visit until discharge or death, assessed up to 12 months
  Assessment of the patient´s peripheral oxygen saturation will be performed at all visits during the acute phase.

CONTACTS AND LOCATIONS:
Overall Officials: Jörg J Vehreschild, Prof., Principal Investigator — Johann Wolfgang Goethe-Universität Frankfurt am Main
Locations (34):
- Germany (34):
  - RWTH Aachen, Aachen
  - University Hospital Augsburg, Augsburg
  - Charité Berlin, Berlin
  - Klinikum Bielefeld, Bielefeld
  - University Hospital Ruhr-University Bochum, Bochum
  - University Hospital Bonn, Bonn
  - University Hospital Cologne, Cologne
  - University Hospital Carl Gustav Carus Dresden, Dresden
  - University Hospital Dusseldorf, Düsseldorf
  - University Hospital Erlangen, Erlangen
  - University Hospital Essen, Essen
  - Johann Wolfgang Goethe University, Frankfurt am Main
  - University Hospital Freiburg, Freiburg im Breisgau
  - University Hospital Göttingen, Göttingen
  - University Hospital Greifswald, Greifswald
  - University Hospital Halle, Halle
  - University Hospital Hamburg-Eppendorf, Hamburg
  - University Hospital MMH Hannover, Hanover
  - University Hospital Heidelberg, Heidelberg
  - University Hospital UKS Homburg, Homburg
  - University Hospital Jena, Jena
  - University Hospital UKSH Schleswig-Holstein, Kiel
  - University Hospital Leipzig, Leipzig
  - University Hospital UKSH Schleswig-Holstein, Lübeck
  - University Hospital Mannheim, Mannheim
  - University Hospital Giessen/Marburg, Marburg
  - University Hospital LMU Munich, Munich
  - University Hospital TUM Munich, Munich
  - University Hospital Münster, Münster
  - Klinikum Oldenburg, Oldenburg
  - University Hospital Regensburg, Regensburg
  - University Hospital Tübingen, Tübingen
  - University Hospital Ulm, Ulm
  - University Hospital Würzburg, Würzburg

IPD SHARING:
Plan to Share IPD: No
Please see use and access conditions according to www.napkon.de

REFERENCES:
- [Derived] Appel KS, Lee CH, Nunes de Miranda SM, Maier D, Reese JP, Anton G, Bahmer T, Ballhausen S, Balzuweit B, Bellinghausen C, Blumentritt A, Brechtel M, Chaplinskaya-Sobol I, Erber J, Fiedler K, Geisler R, Heyder R, Illig T, Kohls M, Kollek J, Krist L, Lorbeer R, Miljukov O, Mitrov L, Nurnberger C, Pape C, Pley C, Schafer C, Schaller J, Schattschneider M, Scherer M, Schulze N, Stahl D, Stubbe HC, Tamminga T, Tebbe JJ, Vehreschild MJGT, Wiedmann S, Vehreschild JJ. A precise performance-based reimbursement model for the multi-centre NAPKON cohorts - development and evaluation. Sci Rep. 2024 Jun 13;14(1):13607. doi: 10.1038/s41598-024-63945-5. PMID 38871878
- [Derived] Hopff SM, Appel KS, Miljukov O, Schneider J, Addo MM, Bals R, Bercker S, Blaschke S, Brohl I, Buchner N, Dashti H, Erber J, Friedrichs A, Geisler R, Gopel S, Hagen M, Hanses F, Jensen BO, Keul M, Krawczyk A, Lorenz-Depiereux B, Meybohm P, Milovanovic M, Mitrov L, Nurnberger C, Obst W, Rommele C, Schafer C, Scheer C, Scherer M, Schmidt J, Seibel K, Sikdar S, Tebbe JJ, Tepasse PR, Thelen P, Vehreschild MJGT, Weismantel C, Vehreschild JJ. Comparison of post-COVID-19 symptoms in patients infected with the SARS-CoV-2 variants delta and omicron-results of the Cross-Sectoral Platform of the German National Pandemic Cohort Network (NAPKON-SUEP). Infection. 2024 Dec;52(6):2253-2267. doi: 10.1007/s15010-024-02270-5. Epub 2024 May 3. PMID 38700656
- [Derived] Appel KS, Nurnberger C, Bahmer T, Forster C, Polidori MC, Kohls M, Kraus T, Hettich-Damm N, Petersen J, Blaschke S, Brohl I, Butzmann J, Dashti H, Deckert J, Dreher M, Fiedler K, Finke C, Geisler R, Hanses F, Hopff SM, Jensen BO, Konik M, Lehnert K, de Miranda SMN, Mitrov L, Miljukov O, Reese JP, Rohde G, Scherer M, Tausche K, Tebbe JJ, Vehreschild JJ, Voit F, Wagner P, Weigl M, Lemhofer C; NAPKON Study Group. Definition of the Post-COVID syndrome using a symptom-based Post-COVID score in a prospective, multi-center, cross-sectoral cohort of the German National Pandemic Cohort Network (NAPKON). Infection. 2024 Oct;52(5):1813-1829. doi: 10.1007/s15010-024-02226-9. Epub 2024 Apr 8. PMID 38587752
- [Derived] Schons M, Pilgram L, Reese JP, Stecher M, Anton G, Appel KS, Bahmer T, Bartschke A, Bellinghausen C, Bernemann I, Brechtel M, Brinkmann F, Brunn C, Dhillon C, Fiessler C, Geisler R, Hamelmann E, Hansch S, Hanses F, Hanss S, Herold S, Heyder R, Hofmann AL, Hopff SM, Horn A, Jakob C, Jiru-Hillmann S, Keil T, Khodamoradi Y, Kohls M, Kraus M, Krefting D, Kunze S, Kurth F, Lieb W, Lippert LJ, Lorbeer R, Lorenz-Depiereux B, Maetzler C, Miljukov O, Nauck M, Pape D, Puntmann V, Reinke L, Rommele C, Rudolph S, Sass J, Schafer C, Schaller J, Schattschneider M, Scheer C, Scherer M, Schmidt S, Schmidt J, Seibel K, Stahl D, Steinbeis F, Stork S, Tauchert M, Tebbe JJ, Thibeault C, Toepfner N, Ungethum K, Vadasz I, Valentin H, Wiedmann S, Zoller T, Nagel E, Krawczak M, von Kalle C, Illig T, Schreiber S, Witzenrath M, Heuschmann P, Vehreschild JJ; NAPKON Research Group. The German National Pandemic Cohort Network (NAPKON): rationale, study design and baseline characteristics. Eur J Epidemiol. 2022 Aug;37(8):849-870. doi: 10.1007/s10654-022-00896-z. Epub 2022 Jul 29. PMID 35904671
- See also: More information on the study and the cross-sectoral platform is provided on the National Pandemic Cohort Network (NAPKON) website. — https://napkon.de/